CLINICAL TRIAL: NCT03949231
Title: A Phase II/III Randomized Trial of Comparison of Survival Benefit of Administration of PD1/PDL1/CTLA4 Inhibitor or Their Combinations Via Hepatic Arterial Infusion Versus Vein for Immunotherapy of Advanced Liver Cancer
Brief Title: Infusion of PD1/PDL1/CTLA4 Inhibitors Via Hepatic Arterial for Immunotherapy of Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZIAICI-008
Record Dates: First submitted 2019-05-13; First posted 2019-05-14 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Liver Cancer
Keywords: Liver Cancer; PD1 antibody; Artery infusion; PDL1 antibody; CTLA4 antibody
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD1/PDL1/CTLA4 inhibitor or their combinations hepatic artery infusion (Experimental): Interventional technique to place microcatheter in hepatic artery to infuse PD1/PDL1/CTLA4 inhibitor or their combinations in 30 minutes.
  Interventions: Drug: PD1/PDL1 inhibitor
- PD1/PDL1/CTLA4 inhibitor or their combinations vein infusion (Experimental): Regular IV infusion of PD1/PDL1/CTLA4 inhibitor or their combinations in 30 minutes.
  Interventions: Drug: PD1/PDL1 inhibitor

INTERVENTIONS:
Drug: PD1/PDL1 inhibitor — Infusion of PD1/PDL1 inhibitor through peripheral vein or hepatic artery.
  Other Names: Administration of PD1/PDL1 inhibitor through vein or interventional technique.

SUMMARY:
This trial was designed to investigate the survival outcomes, response rates, and safety of patients with Barcelona-Clinical Hepatocellular Carcinoma (BCLC)-C-stage liver cancer by hepatic artery versus vein infusion of PD1/PDL1/CTLA4 inhibitor or their combinations.

DETAILED DESCRIPTION:
Liver cancer is the fifth most common malignancy worldwide, but the mortality rate ranks third. China has a large population base, with more than 400,000 new cases each year, and more than half of the world's new liver cancer and deaths. More than 70% of liver cancer patients in China are diagnosed at mid-to-late stage and have lost the chance of surgery. Only 10%-15% of newly diagnosed patients can undergo radical resection, and the recurrence rate after 5 years is as high as 50%-80%. So far, sorafenib is still the only standard treatment that can prolong the overall survival of advanced hepatocellular carcinoma. SHARP's latest research shows that sorafenib can only extend patients with advanced liver cancer for 2.8 months, and many adverse reactions; regofenib can be used in patients with advanced liver cancer after taking sorafenib resistance, but the overall efficiency is still low. It is difficult to be widely used in patients with advanced liver cancer, and more alternative therapies are urgently needed.

PD1/PDL1 inhibitor is widely used in treatment of various cancers in China now. The hepatic arterial chemotherapy infusion for advanced liver cancer, through the "first pass effect" of drug treatment, can significantly increase the local drug concentration of the tumor, improve the efficacy, reduce systemic adverse reactions, meanwhile Folfox regimen has been confirmed by the hepatic arterial chemotherapy infusion program. To the investigator's knowledge, no studies have been developed on the survival benefit of hepatic arterial infusion of immunotherapeutic agents in patients with advanced liver cancer. This phase III clinical trial was designed to compare the effects of PD1/PDL1/CTLA4 inhibitor or their combinations via IA and IV on the survival benefit of patients with advanced liver cancer, including ORR, DCR, median survival time, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Cytohistological confirmation is required for diagnosis of HCC.、
2. Signed informed consent before recruiting
3. Age between 18 to 80 years with estimated survival over 3 months.
4. Child-Pugh class A or B/Child score > 7; ECOG score < 2
5. Tolerable coagulation function or reversible coagulation disorders
6. Laboratory examination test within 7 days prior to procedure: WBC≥3.0×10E9/L; Hb≥90g/L； PLT ≥50×10E9/L；INR < 2.3 or PT < 6 seconds above control；Cr ≤ 145.5 umul/L；Albumin > 28 g/L；Total bilirubin < 51 μmol/L
7. At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.
8. Patients with advanced (unresectable and/or metastatic, stage C based on Barcelona-Clinic Liver Cancer [BCLC] staging classification) hepatocellular carcinoma which would not be suitable for treatment with loco-regional therapies or have progressed following locoregional therapy such as surgical resection, percutaneous hepatic arterial embolization, radiofrequency ablation, and percutaneous interventional therapy.
9. Birth control.
10. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Patients participated in clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
2. Patients accompany by ascites, hepatic encephalopathy and esophageal and gastric varices bleeding;
3. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
4. Patients accompanied with other tumors or past medical history of malignancy;
5. Pregnant or lactating patients, all patients participating in this trial must adopt appropriate birth control measures during treatment;
6. Patients have poor compliance.

   Any contraindications for hepatic arterial infusion procedure:

   A.Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).

   B.Renal failure / insufficiency requiring hemo-or peritoneal dialysis. C.Known severe atheromatosis. D.Known uncontrolled blood hypertension (> 160/100 mm/Hg).
7. Patients have the past history of liver cancer treatment, such as transplantation, resection, radiotherapy, chemotherapy and so on;
8. Allergic to adriamycin chemotherapy drugs，contrast agent and lipiodol;
9. Any agents which could affect the absorption or pharmacokinetics of the study drugs
10. Subjects unable to suffer the discomfort of the HAI procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2038-01-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will occur every 12 weeks (±1 month) until death or withdrawal of consent from the study.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per mRECIST) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Adverse event rate | 2 years
  Adverse event rate will be defined as the rate of patients who developed adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Lian, MD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University; Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong, China